CLINICAL TRIAL: NCT07022327
Title: IMPACT Study: Intervention Monitoring for Pancreatitis in an Adolescent Undergoing Clinical Treatment
Brief Title: Ivacaftor Impact in an Adolescent Without a Cystic Fibrosis-Associated CFTR (Cystic Fibrosis Transmembrane Conductance Regulator) Mutation for Chronic Pancreatitis: Single-Patient Study Tracking Flare Frequency and Health Data Compared to Historical Records.
Acronym: IMPACT
Status: Active, not recruiting | Type: Observational
Sponsor: Mission: Cure (Other)
Responsible Party: Sponsor
Other Study IDs: N1-IVAC-01; 20251496 (Other: WCG)
Record Dates: First submitted 2025-06-07; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — ivacaftor; Magnesium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Ivacaftor 150 MG (milligrams) — Ivacaftor is a CFTR potentiator approved for the treatment of cystic fibrosis in patients with specific gating mutations. In this observational, single-patient study, Ivacaftor is being used off-label in an adolescent without a cystic fibrosis-associated CFTR mutation to evaluate its potential impact on chronic pancreatitis. The intervention is not assigned by the study team but is part of the participant's ongoing medical care. The study monitors clinical outcomes and wearable health data over a 12-month period.

SUMMARY:
The goal of this observational study is to learn about the long-term effects of Ivacaftor in an adolescent without a cystic fibrosis-associated CFTR mutation who is taking Ivacaftor to treat chronic pancreatitis. The main question it aims to answer is:

Does Ivacaftor reduce the frequency or severity of acute pancreatitis episodes in this adolescent compared to their historical medical data?

The participant, who is already taking Ivacaftor as part of their medical care, will be monitored over the course of 12 months. Flare frequency, hospitalizations, and wellness data will be tracked through caregiver reports, lab data, and physiological data collected from a wearable health monitoring device (Apple Watch).

ELIGIBILITY:
Inclusion Criteria:

The subject has been diagnosed with recurrent acute pancreatitis or chronic pancreatitis and a clinical decision has been made to treat the subject with one or more FDA-approved therapies, which may be being used off-label) to treat or prevent pancreatitis symptoms.

Exclusion Criteria:

Participant has a known cystic fibrosis-associated CFTR mutation that would qualify them for standard Ivacaftor use.

Participant is unable to tolerate Ivacaftor due to prior adverse reactions.

Participant has severe liver dysfunction or baseline liver enzyme elevations that contraindicate Ivacaftor use, as determined by the treating physician.

Participant or parent/guardian is unwilling to comply with study procedures, including regular follow-up and data sharing.

Any other medical or psychological condition, in the judgment of the treating physician or counselor, that would make participation unsafe or not in the best interest of the participant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of a single adolescent under the age of 16 with a clinical diagnosis of chronic pancreatitis, who has experienced recurrent acute-on-chronic pancreatitis episodes despite standard treatments. The participant does not carry a cystic fibrosis-associated CFTR mutation associated with Cystic Fibrosis and is under the ongoing care of a multidisciplinary team. This individual was selected for observation based on persistent disease burden, lack of response to conventional therapies, and medical decision-making that included initiating off-label Ivacaftor use as part of the participant's clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Time Between Acute Pancreatitis Episodes While on Ivacaftor | 12 months
  The number of days between clinically confirmed acute pancreatitis attacks during the 12-month Ivacaftor treatment period, compared to historical pre-treatment intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Schork, PhD, Principal Investigator — Net.bio
Locations (1):
- Mission: Cure, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT07022327/Prot_SAP_000.pdf